CLINICAL TRIAL: NCT01070394
Title: Evaluation of Pharmacokinetics and Profile of Clinical Response of Subacute Lisdexamfetamine Dimesylate (Vyvanse) Treatment vs. Clinical Response to Subacute Immediate Release Mixed Amphetamine Salt Therapy in Adult ADHD
Brief Title: Effectiveness and Duration of Effect of Open Treatment in Attention Deficit Hyperactivity Disorder (ADHD) Patients Treated With Lisdexamfetamine Dimesylate(Vyvanse)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-00510
Record Dates: First submitted 2010-02-16; First posted 2010-02-18 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Lisdexamfetamine Dimesylate; Amphetamine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LDX Treatment (Experimental): Eligible participants received 12 weeks of open-label treatment. Those on treatment prior to baseline underwent a 7-day (for amphetamine or methylphenidate) or 28-day (for atomoxetine or other medications) washout period prior to initiating LDX treatment. The starting dose was 30mg/day, which could be titrated up by 20mg/day during visits 2-6 (for a maximum dose of 70mg/day). At discretion of investigator, the dose could be down-titrated by 20mg/day during visits 4-6. Once the dose was optimized (after visit 6), the dose was maintained for 8 weeks.
  Interventions: Drug: LDX Treatment

INTERVENTIONS:
Drug: LDX Treatment — 30 mg, 50mg, or 70 mg. Oral capsule, once a day, for 12 weeks.
  Other Names: Vyvanse

SUMMARY:
The purpose of this study is to examine the effectiveness and length of effect of Vyvanse on lessening Attention-Deficit/Hyperactivity Disorder symptoms in adults. The study will also investigate the safety and tolerability of Vyvanse in adults with ADHD.

DETAILED DESCRIPTION:
Protocol Summary:

Effectiveness and Duration of Effect of Open Treatment in Adult ADHD Patients Treated with Lisdexamfetamine Dimesylate- LDX (Vyvanse)

The primary objective of this study is to evaluate the effectiveness and duration of effect of LDX for the treatment of ADHD symptoms in adults. The study will be a 12-week open label extension with 25 adult participants who completed a cross-over study of adherence/efficacy of Adderall Immediate Release (IR) vs. Adderall Extended Release (XR).

The secondary objective is to provide information regarding tolerability, dosing and titration of LDX in the adult population with ADHD.

An additional fifteen participants will be recruited using advertising and previous Mental Health and Addictive Behaviour Research Program (MHADRP) studies will be offered treatment with LDX. All participants will be diagnosed with ADHD using the Adult Clinician Diagnostic Scale (ACDS). We will be collecting demographic information, administering the Scheduled Clinical Interview for DSM Disorders (SCID), collecting medical history, previous drug therapy, and the participant will have a physical with the physician. A coordinator will give an electrocardiogram (ECG), and collect a blood sample for blood chemistry and hematology.

Schedule of Events: Vyvanse Extension Screening Visit

* Consent
* Demographics (needs to be added?)
* Physical
* Medical history (needs to be added?)
* Previous drug therapy
* Vitals (Blood Pressure-BP, Heart Rate-HR, Respiration, weight)
* Urine Drug screen
* Urine pregnancy test
* ECG
* Blood sample
* SCID
* ACDS

Visits at week 0,1,2,3,4,6,8,10,12 (every visit)

* ADHD-Rating Scale (ADHD-RS)
* Adult ADHD Self-Report Scale (ASRS)
* Clinical Global Impression (CGI)
* Vitals
* Pill count
* Adverse Events (AE)/ Concomitant Medications (CM)

Visits at week 0,1,4,6,12 also administer

* Adult ADHD Medication Rebound Scale (AMRS) (AM/PM)
* Adult ADHD Medication Smoothness of Effect Scale (AMSES) (AM/PM)
* Wender-Reimherr Adult Attention Deficit Disorder Scale (WRAADS) (AM/PM)

First 4 weeks of treatment is a dose adjustment period (30-70 mg po qAM), after those 4 weeks established dose is remained for remaining 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of consent, are between the ages of 18-55, inclusive.
2. Meet DSM-IV criteria for ADHD as assessed by the Adult ADHD Clinician Diagnostic Scale (ACDS) v1.2.
3. Female participants of childbearing potential must test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use a reliable method of birth control during the study. Females of childbearing potential are defined as women not surgically sterilized and are between menarche and 2 years post-menopause.
4. Must have a satisfactory medical assessment with no clinically significant abnormalities as determined by medical history, physical exam, ECG, and clinical laboratory testing.
5. Must be able to swallow capsules.
6. Must be able to begin the daily dose of study medication in the morning.
7. Must be off all ADHD therapies for one week (psychostimulants) and three weeks (non-stimulants).
8. In the opinion of the investigator, the subject must understand and be able, willing and likely to fully comply with the study procedures and restrictions.
9. Must have given signed and dated informed consent in accordance with Good Clinical Practice (GCP) Guidelines.

Exclusion Criteria:

1. Participants with a positive urine drug result at Screening.
2. Anyone who meets current DSM-IV-TR criteria for alcohol or any non-alcohol substance abuse or dependence disorder (excluding nicotine).
3. Participants with controlled depressive or anxiety disorders may not participate if, in the opinion of the Principal Investigator, their medications will interfere with safety or efficacy assessments.
4. Participants with any concurrent chronic or acute illness or unstable medical condition that could, in the opinion of the study physician, confound the results of safety assessments, increase risk to the subject or lead to difficulty complying with the protocol.
5. Participants with hypertension at screening, indicated by a blood pressure reading of 135/90 and heart rate above 120bmp.
6. Female participants of childbearing potential who test positive for pregnancy at the time of enrollment based on a urine pregnancy test, or who do not agree to use a reliable method of birth control during the study. Females of childbearing potential are defined as women not surgically sterilized and are between menarche and 2 years post-menopause.
7. Participants who work the night shift or another schedule that would preclude beginning the daily dose of study medication in the morning.
8. Participants who in the investigator's opinion meet any of the exclusionary criteria specified on the FDA label of Vyvanse.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lenard Adler, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Adler LA, Alperin S, Leon T, Faraone S. Clinical effects of lisdexamfetamine and mixed amphetamine salts immediate release in adult ADHD: results of a crossover design clinical trial. Postgrad Med. 2014 Sep;126(5):17-24. doi: 10.3810/pgm.2014.09.2796. PMID 25295646
- [Derived] Mattingly GW, Weisler RH, Young J, Adeyi B, Dirks B, Babcock T, Lasser R, Scheckner B, Goodman DW. Clinical response and symptomatic remission in short- and long-term trials of lisdexamfetamine dimesylate in adults with attention-deficit/hyperactivity disorder. BMC Psychiatry. 2013 Jan 29;13:39. doi: 10.1186/1471-244X-13-39. PMID 23356790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first 25 participants enrolled consisted of adults who had recently completed a randomized, cross-over, open label study (MAS Adherence Study) that examined adherence to ADHD treatment with MAS IR vs. MAS XR. An additional 15 adults were recruited from local advertising and from the pool of participants at the MHADRP at the NYU SoM.
Pre-assignment Details: Participants taking prohibited concomitant medications, including ADHD medications, will be required to washout of their medication during the screening phase.The washout period will be one week for psychostimulants and three weeks for non-stimulants.
Groups:
- Overall Study: Lisdexamfetamine Treatment: The treatment arm will receive 12 weeks of Lisdexamfetamine Dimesylate-LDX treatment. At baseline, participants were initiated on LDX at a dose of 30 mg/day and began a 4-week dose optimization phase with weekly clinic visits. The dose optimization phase was followed by an 8-week dose maintenance phase, which included clinic visits every 2 weeks for the assessment of safety and efficacy. At visits 3-6, the dose of LDX was increased by 20 mg/day until an optimal dose or the maximum dose of 80 mg/day was reached. An optimal dose was determined by clinical efficacy, defined as a >= 30% reduction in the baseline ADHD Rating Scale, and tolerability. At the discretion of the investigator, the dose could be down-titrated by 20 mg/day at visits 4-6. When an optimal dose was reached, the participant remained at this level for the duration of the study.
Period: Overall Study
Arm/Group | Overall Study: Lisdexamfetamine Treatment
Started | 40
Completed | 33
Not Completed | 7
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Eligibility was determined by meeting all inclusion criteria and not meeting any of the exclusion criteria. Of the 40 who initially enrolled, 33 completed the full treatment.
Groups:
- LDX Treatment: Prospective participants will be evaluated for ADHD and study inclusion/exclusion criteria. Eligible participants will begin open-label lisdexamfetamine dimesylate for 12 weeks. Those who were able to complete all 12 weeks of the treatment were evaluated for data purposes.
Arm/Group | LDX Treatment
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 21
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 21
  Black or African-American | 5
  Hispanic | 2
  Asian | 3
  Other/Mixed Ethnicity | 2

OUTCOME MEASURES:

1. Secondary Outcome: Change in Symptom Rebound Score Using the Adult ADHD Medication Rebound Scale (AMRS).
Description: To evaluate the symptom rebound throughout a single day (assessed via the AMRS) with LDX treatment. Scoring on the AMRS based on 38 items, each scored 0 (None), 1 (Mild), 2 (Moderate), 3 (Severe). The lowest scored units on a scale for 1 individual is 0, the highest 114. The scores reported below are Mean scores for 33 patients analyzed.
Time Frame: Week 0 to Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Overall Study: Eligible participants received 12 weeks of open-label treatment. Those on treatment prior to baseline underwent a 7-day (for amphetamine or methylphenidate) or 28-day (for atomoxetine or other medications) washout period prior to initiating LDX treatment. The starting dose was 30mg/day, which could be titrated up by 20mg/day during visits 2-6 (for a maximum dose of 70mg/day). At discretion of investigator, the dose could be down-titrated by 20mg/day during visits 4-6. Once the dose was optimized (after visit 6), the dose was maintained for 8 weeks.
  LDX Treatment: 30 mg, 50mg, or 70 mg. Oral capsule, once a day, for 12 weeks.
Arm/Group | Overall Study
Number analyzed (Participants) | 33
units on a scale
  In Clinic | 27.99 (4.17)
  Evening | 26.9 (5.29)
Statistical Analysis 1: Comparison: Overall Study; Test type: Superiority or Other; p < .001, GEE regression model; Generalized Estimating Equation (GEE)

2. Secondary Outcome: Change in Measure of Smoothness of Effect Using Adult ADHD Medications Smoothness of Effect Scale (AMSES)
Description: The Adult ADHD Medication Smoothness of Effect Scale (AMSES) is a 6-item, frequency-based, self-report scale that was recently developed to assess the consistency and duration of effect of ADHD medication throughout the day. The AMSES compares the effectiveness of ADHD medication shortly after dosing with the effectiveness later in the day. Respondents are asked to rate how frequently the effective-ness of their medication was the same 2 hr post-dose as it was 4, 6, 8, 10, and 12 hr post-dose on a 0 to 4 scale (0 = never, 1 = rarel, 2 = sometimes, 3 = often, 4 = very often). In addition, respondents rate how frequently the delivery of their medication was consistent and smooth throughout the day on a visual analog scale ranging from 0 (never) to 100 (very often).
Time Frame: Visits 0 and 12
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Overall Study: The treatment arm will receive 12 weeks of Lisdexamfetamine Dimesylate-LDX treatment. At baseline, participants were initiated on LDX at a dose of 30 mg/day and began a 4-week dose optimization phase with weekly clinic visits. The dose optimization phase was followed by an 8-week dose maintenance phase, which included clinic visits every 2 weeks for the assessment of safety and efficacy. At visits 3-6, the dose of LDX was increased by 20 mg/day until an optimal dose or the maximum dose of 80 mg/day was reached. An optimal dose was determined by clinical efficacy, defined as a >= 30% reduction in the baseline ADHD Rating Scale, and tolerability. At the discretion of the investigator, the dose could be down-titrated by 20 mg/day at visits 4-6. When an optimal dose was reached, the participant remained at this level for the duration of the study.
Arm/Group | Overall Study
Number analyzed (Participants) | 33
units on a scale
  In Clinic | 1.31 (3.70)
  Evening | -3.34 (3.47)
Statistical Analysis 1: Comparison: Overall Study; Test type: Superiority or Other; p = .569, GEE regression model; Generalized Estimating Equation (GEE)
Statistical Analysis 2: Comparison: Overall Study; The following p-value is for AMSES In-Clinic, a subset of the overall AMSES; Test type: Superiority or Other; p = .827, Generalized Estimating Equation
Statistical Analysis 3: Comparison: Overall Study; The following p-value is for AMSES, Evening, a subset of the AMSES; Test type: Superiority or Other; p = .569, Generalized Estimating Equation

3. Secondary Outcome: Correlation Between AMRS (In Clinic) and ADHD-RS
Description: To correlate symptom rebound through a single day (assessed via the AMRS) with a global (ADHD-RS) measure of efficacy of LDX treatment. AMRS and ADHD-RD scores obtained on Day 0 and Day 12 will be correlated. The Pearson's correlation coefficients for the In-Clinic assessment will be presented for Visits 0 and 12.
Time Frame: Visits 0 and 12
Measure: Number; unit: Pearson's correlation coefficient
Groups:
- Treatment Arm: The treatment arm will receive 12 weeks of Lisdexamfetamine Dimesylate-LDX treatment. At baseline, participants were initiated on LDX at a dose of 30 mg/day and began a 4-week dose optimization phase with weekly clinic visits. The dose optimization phase was followed by an 8-week dose maintenance phase, which included clinic visits every 2 weeks for the assessment of safety and efficacy. At visits 3-6, the dose of LDX was increased by 20 mg/day until an optimal dose or the maximum dose of 80 mg/day was reached. An optimal dose was determined by clinical efficacy, defined as a >= 30% reduction in the baseline ADHD Rating Scale, and tolerability. At the discretion of the investigator, the dose could be down-titrated by 20 mg/day at visits 4-6. When an optimal dose was reached, the participant remained at this level for the duration of the study.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 33
Pearson's correlation coefficient | .66
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Superiority or Other; p = .001, GEE regression model; Generalized Estimating Equation (GEE)

4. Secondary Outcome: Change in Correlation Between AMRS and TASS
Description: To correlate symptom rebound through a single day (assessed via the AMRS) with a time-sensitive (TASS) measure of efficacy of LDX treatment. A Pearson's correlation coefficient will be presented. AMRS and TASS scores obtained on Day 0 and Day 12 will be correlated. The Pearson's correlation coefficients for the In-Clinic assessment will be presented for Visits 0 and 12.
Time Frame: Visits 0 and 12
Measure: Number; unit: Pearson's correlation coefficient
Arm/Group | Overall Study
Number analyzed (Participants) | 33
Pearson's correlation coefficient
  In Clinic | .96
  Evening | .96
Statistical Analysis 1: Comparison: Overall Study; Test type: Superiority or Other; p < .001, GEE regression model

5. Secondary Outcome: Correlation Between In-Clinic AMRS and ASRS v.1.1 Symptom Checklist
Description: To correlate symptom rebound through a single day (assessed via the AMRS) with a self assessment of ADHD Symptoms. A Pearson's correlation coefficient will be presented. AMRS and self assessment of ADHD scores obtained on Day 0 and Day 12 will be correlated. The Pearson's correlation coefficients for the In-Clinic assessment will be presented for Visits 0 and 12.
Time Frame: Baseline to Week 12
Measure: Number; unit: Pearson's correlation coefficient
Arm/Group | Overall Study
Number analyzed (Participants) | 33
Pearson's correlation coefficient | .83
Statistical Analysis 1: Comparison: Overall Study; Test type: Superiority or Other; p < .0001, GEE regression model; Generalized Estimating Equation (GEE)

6. Primary Outcome: Attention Deficit Hyperactivity Disorder- Rating Scale (ADHS-RS)
Description: The ADHD-RS with adult ADHD prompts is a semi-structured scale that consists of 18 items that directly correspond to the 18 DSM-IV symptoms of ADHD, and is designed to assess current symptomatology19.
  Each item is scored on a 4-point scale ranging from 0 (none) to 3 (severe).Each item on the 18-item measure is scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms), yielding a possible total score of 0-54. A score of 0-16 means "Unlikely to have ADHD"; a score of 17-23 "Likely to Have ADHD" ; 24 or greater-Highly Likely to have ADHD
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Study
Number analyzed (Participants) | 33
units on a scale | 13.9 (2.31)
Statistical Analysis 1: Comparison: Overall Study; Test type: Superiority or Other; p = 0.001, GEE regression model; Generalized Estimating Equation (GEE)

7. Secondary Outcome: Psychometric Validation of AMRS
Description: To perform secondary psychometric validations of the AMRS using Cronbach's alpha coefficients.
Time Frame: Weeks 0-12
Measure: Number; unit: Cronbach's alpha coefficients
Arm/Group | Overall Study
Number analyzed (Participants) | 33
Cronbach's alpha coefficients
  In Clinic | .99
  Evening | .97

8. Secondary Outcome: Psychometric Validation of AMSES
Description: To perform secondary psychometric validations of the AMSES using Cronbach's alpha coefficients.
Time Frame: Weeks 0-12
Measure: Number; unit: Cronbach's alpha coefficients
Arm/Group | Overall Study
Number analyzed (Participants) | 33
Cronbach's alpha coefficients
  In Clinic | .92
  Evening | .87

ADVERSE EVENTS:
Groups:
- LDX Treatment: The treatment arm will receive 12 weeks of Lisdexamfetamine Dimesylate-LDX treatment. At baseline, participants were initiated on LDX at a dose of 30 mg/day and began a 4-week dose optimization phase with weekly clinic visits. The dose optimization phase was followed by an 8-week dose maintenance phase, which included clinic visits every 2 weeks for the assessment of safety and efficacy. At visits 3-6, the dose of LDX was increased by 20 mg/day until an optimal dose or the maximum dose of 80 mg/day was reached. An optimal dose was determined by clinical efficacy, defined as a >= 30% reduction in the baseline ADHD Rating Scale, and tolerability. At the discretion of the investigator, the dose could be down-titrated by 20 mg/day at visits 4-6. When an optimal dose was reached, the participant remained at this level for the duration of the study.
Arm/Group | LDX Treatment
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 33/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LDX Treatment (N=40)
Insomnia (General disorders) | 32 (34)
Headache (Vascular disorders) | 21 (22)
Loss of Appetite (Gastrointestinal disorders) | 21 (21)
Dry Mouth (General disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No